CLINICAL TRIAL: NCT01741350
Title: Testing a Community-Friendly Risk Reduction Intervention for Injection Drug Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); APT Foundation, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H06-215; 1R01DA022122-01A1 (NIH)
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Results first posted 2014-02-27 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-01

CONDITIONS: HIV; Opioid Dependence
Keywords: Methadone-maintenance; HIV; Risk behavior; Injection drug use; Condom use; Health care participation; Opioid replacement therapy
MeSH Terms: conditions — Opioid-Related Disorders; Risk-Taking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CHRP Group (Experimental): Patients assigned to Community-friendly Health Recovery Program (CHRP) will receive a weekly HIV risk reduction group level intervention led by two facilitators trained and supervised by the PI, a licensed clinical psychologist. The CHRP intervention is a substantially shortened version of the comprehensive Holistic Health Recovery Program (HHRP)-based interventions that have been identified as demonstrating evidence of effectiveness in two randomized clinical trials. The CHRP, which includes four 50-minute groups (1 group per week), will contain only content that relates explicitly to drug- or sex-related HIV risk reduction. Participants in both conditions will receive routine clinical services (i.e., daily methadone and case management).
  Interventions: Behavioral: Community-friendly Health Recovery Program
- Control Condition (Active Comparator): The time-and-attention-matched control condition for the proposed research will be a time and contact-matched, non-contaminating support group for individuals in recovery modeled after similar groups offered in the community. There will be no overlap between the content of the comparison intervention and experimental intervention although the basic structure will be the same. Thus, each participant will be asked to attend four 50-minute weekly group sessions led by two trained facilitators. Participants in both conditions will receive routine clinical services (i.e., daily methadone and case management).
  Interventions: Behavioral: Time-and-Attention-Matched Control Condition

INTERVENTIONS:
Behavioral: Community-friendly Health Recovery Program — Four weekly HIV risk-reduction groups and routine clinical services (i.e., daily methadone and case management).
  Other Names: CHRP
  Arms: CHRP Group
Behavioral: Time-and-Attention-Matched Control Condition — Four weekly support groups and routine clinical services (i.e., daily methadone and case management).
  Arms: Control Condition

SUMMARY:
To conduct a randomized clinical trial (RCT) of a community-friendly behavioral intervention designed to reduce HIV risk behavior among injection drug users (IDUs) in drug treatment by comparing risk-behavior outcomes of four weekly intervention sessions with a time-and-attention-matched control condition.

DETAILED DESCRIPTION:
This research study will test the effects of CHRP, a community-friendly risk reduction intervention, which is based on the Information-Motivation-Behavioral Skills model of health behavior change (IMB; Fisher & Fisher, 1992), and, thus, is designed to enhance knowledge, motivation, and behavior skills for reducing drug- and sex-related HIV risk behaviors. Outcomes assessed will include urine toxicology screens, self-reported HIV drug- and sex-related HIV risk behavior, HIV/AIDS knowledge, risk reduction motivation, and risk reduction behavioral skills.

To measure the effects of CHRP, the investigators are proposing a two-condition (standard of care plus the CHRP intervention vs. standard of care plus a time-and-attention matched control condition) randomized design, balancing for participant gender. The investigators will assess participants at baseline, immediately post-intervention (i.e., at 4 weeks), and at 3-, 6-, and 12-month measurement points following the intervention. This assessment approach will allow the investigators to examine the trajectory of HIV risk reduction change including the decay or emergence of intervention effects.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Opioid-dependent and seeking methadone maintenance treatment
* Report drug- or sex-related HIV risk behavior in previous 6 months
* Able to read and understand the questionnaires, Audio Computer Assisted Self Interview (ACASI), and consent form
* Available for the full duration of the study with no anticipated circumstances impeding participation (e.g., jail term)
* Not actively suicidal, homicidal, or psychotic as assessed by trained research staff under the supervision of a licensed clinical psychologist

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2006-09; Primary Completion 2011-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Copenhaver, Ph.D., Principal Investigator — University of Connecticut
Locations (1):
- APT Foundation, New Haven, Connecticut, United States

REFERENCES:
- [Background] Fisher JD, Fisher WA. Changing AIDS-risk behavior. Psychol Bull. 1992 May;111(3):455-74. doi: 10.1037/0033-2909.111.3.455. PMID 1594721
- [Background] Institute of Medicine (US) Committee on Community-Based Drug Treatment; Lamb S, Greenlick MR, McCarty D, editors. Bridging the Gap between Practice and Research: Forging Partnerships with Community-Based Drug and Alcohol Treatment. Washington (DC): National Academies Press (US); 1998. Available from http://www.ncbi.nlm.nih.gov/books/NBK230402/ PMID 25101381
- See also: Center for Health, Intervention, and Prevention — http://www.chip.uconn.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 648 participants were screened from March 2007 through August 2010 from a methadone maintenance program in New Haven, Connecticut.
Pre-assignment Details: 292 participants did not meet the study's inclusion criteria, 36 participants missed the initial interview appointment, and 16 participants were ineligible due to already being enrolled in another study.
Groups:
- CHRP Group: Patients assigned to Community-friendly Health Recovery Program (CHRP) will receive a weekly HIV risk reduction group level intervention led by two facilitators trained and supervised by the PI, a licensed clinical psychologist. The CHRP intervention is a substantially shortened version of the comprehensive Holistic Health Recovery Program (HHRP)-based interventions that have been identified as demonstrating evidence of effectiveness in two randomized clinical trials. The CHRP, which includes four 50-minute groups (1 group per week), will contain only content that relates explicitly to drug- or sex-related HIV risk reduction. Participants in both conditions will receive routine clinical services (i.e., daily methadone and case management).
  Community-friendly Health Recovery Program : Four weekly HIV risk-reduction groups and routine clinical services (i.e., daily methadone and case management).
- Control Condition: The time-and-attention-matched control condition for the proposed research will be a time and contact-matched, non-contaminating support group for individuals in recovery modeled after similar groups offered in the community. There will be no overlap between the content of the comparison intervention and experimental intervention although the basic structure will be the same. Thus, each participant will be asked to attend four 50-minute weekly group sessions led by two trained facilitators. Participants in both conditions will receive routine clinical services (i.e., daily methadone and case management).
  Time-and-Attention-Matched Control Condition : Four weekly support groups and routine clinical services (i.e., daily methadone and case management).
Period: Study Intervention
Arm/Group | CHRP Group | Control Condition
Started | 149 | 155
Completed | 149 | 155
Not Completed | 0 | 0
Period: Post Intervention Assessment (at Week 4)
Arm/Group | CHRP Group | Control Condition
Started | 149 | 155
Completed | 135 | 141
Not Completed | 14 | 14
Period: 3-Month Follow-up Assessment
Arm/Group | CHRP Group | Control Condition
Started | 135 | 141
Completed | 129 | 119
Not Completed | 6 | 22
Period: 6-Month Follow-up Assessment
Arm/Group | CHRP Group | Control Condition
Started | 129 | 119
Completed | 114 | 111
Not Completed | 15 | 8
Period: 12-Month Follow-up Assessment
Arm/Group | CHRP Group | Control Condition
Started | 114 | 111
Completed | 111 | 109
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Population: Only participants who completed all 5 time points on drug-risk reduction knowledge and personal motivation for safer drug use were included in the analysis (i.e., 95 participants for the intervention group and 90 participants for the control group). For all other variables, the participants analyzed for the two groups were 97 and 92, respectively.
Groups:
- Total: Total of all reporting groups
Arm/Group | CHRP Group | Control Condition | Total
Number analyzed (Participants) | 149 | 155 | 304
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 149 | 155 | 304
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.26 (9.939) | 33.50 (9.141) | 33.87 (9.532)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 81 | 157
  Male | 73 | 74 | 147
Region of Enrollment [Number; unit: participants]
  United States | 149 | 155 | 304

OUTCOME MEASURES:

1. Primary Outcome: Demonstrated Drug Risk Reduction Skills (0-100%)
Description: Participants' HIV risk reduction skills were assessed by having participants demonstrate the steps necessary to properly clean a needle/syringe.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: Percentage of correct steps
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
Percentage of correct steps | 40.60 (1.99) | 42.75 (2.09)

2. Primary Outcome: Demonstrated Drug Risk Reduction Skills (0-100%)
Description: as for outcome 1
Time Frame: Immediately Post-Intervention, at 4 weeks
Measure: Mean (Standard Error); unit: Percentage of correct steps
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
Percentage of correct steps | 76.37 (2.03) | 53.11 (2.14)

3. Primary Outcome: Demonstrated Drug Risk Reduction Skills (0-100%)
Description: as for outcome 1
Time Frame: 3-month follow up
Measure: Mean (Standard Error); unit: Percentage of correct steps
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
Percentage of correct steps | 69.59 (2.04) | 60.34 (2.15)

4. Primary Outcome: Demonstrated Drug Risk Reduction Skills (0-100%)
Description: as for outcome 1
Time Frame: 6-month follow up
Measure: Mean (Standard Error); unit: Percentage of correct steps
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
Percentage of correct steps | 74.12 (1.97) | 63.12 (2.07)

5. Primary Outcome: Demonstrated Drug Risk Reduction Skills (0-100%)
Description: as for outcome 1
Time Frame: 12-month follow up
Measure: Mean (Standard Error); unit: Percentage of correct steps
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
Percentage of correct steps | 72.61 (1.91) | 63.63 (2.01)

6. Primary Outcome: Safer Drug Use (0-4)
Description: Participants completed a self-reported assessment that asks about IV-sharing behavior and were assessed on a scale of 0-4, with higher scores indicating safer drug use.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 3.25 (0.10) | 3.39 (0.10)

7. Primary Outcome: Safer Drug Use (0-4)
Description: as for outcome 6
Time Frame: Immediately Post-Intervention, at 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 3.78 (0.06) | 3.79 (0.06)

8. Primary Outcome: Safer Drug Use (0-4)
Description: as for outcome 6
Time Frame: 3-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 3.83 (0.05) | 3.81 (0.05)

9. Primary Outcome: Safer Drug Use (0-4)
Description: as for outcome 6
Time Frame: 6-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 3.84 (0.05) | 3.77 (0.05)

10. Primary Outcome: Safer Drug Use (0-4)
Description: as for outcome 6
Time Frame: 12-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 92 | 92
units on a scale | 3.87 (0.05) | 3.85 (0.05)

11. Primary Outcome: Drug-related HIV-risk Reduction Knowledge (0-1)
Description: Participants completed an assessment that covers information about drug-related HIV-risk reduction (e.g.,"If an HIV+ person shared needles with another HIV+ person, they don't need to clean the needles") and were rated on a scale of 0 to 1 (higher values representing greater risk reduction knowledge).
Time Frame: Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 95 | 90
units on a scale | 0.96 (0.02) | 1.00 (0.02)

12. Primary Outcome: Drug-related HIV-risk Reduction Knowledge (0-1)
Description: as for outcome 11
Time Frame: Immediately Post-Intervention, at 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 95 | 90
units on a scale | 1.00 (0.01) | 0.98 (0.01)

13. Primary Outcome: Drug-related HIV-risk Reduction Knowledge (0-1)
Description: as for outcome 11
Time Frame: 3-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 95 | 90
units on a scale | 1.00 (0.01) | 0.96 (0.01)

14. Primary Outcome: Drug-related HIV-risk Reduction Knowledge (0-1)
Description: as for outcome 11
Time Frame: 6-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 95 | 90
units on a scale | 0.96 (0.02) | 0.99 (0.02)

15. Primary Outcome: Drug-related HIV-risk Reduction Knowledge (0-1)
Description: Participants completed an assessment that covers information about drug-related HIV-risk reduction (e.g.,"If an HIV+ person shared needles with another HIV+ person, they don't need to clean the needles").
Time Frame: 12-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 95 | 90
units on a scale | 0.98 (0.02) | 0.96 (0.02)

16. Primary Outcome: Personal Motivation to Reduce Drug-related HIV-Risk Behavior (1-5)
Description: Participants completed a questionnaire assessing their personal motivation to reduce HIV risk behavior (e.g., "I plan to always use clean needles if I shoot up drugs during the next six months") and rated on a scale of 1 to 5, with higher scores indicating stronger motivation to reduce HIV-risk behavior.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 95 | 90
units on a scale | 4.79 (0.05) | 4.85 (0.05)

17. Primary Outcome: Personal Motivation to Reduce Drug-related HIV-Risk Behavior (1-5)
Description: as for outcome 16
Time Frame: Immediately Post-Intervention, at 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 95 | 90
units on a scale | 4.91 (0.05) | 4.83 (0.05)

18. Primary Outcome: Personal Motivation to Reduce Drug-related HIV-Risk Behavior (1-5)
Description: as for outcome 16
Time Frame: 3-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 95 | 90
units on a scale | 4.87 (0.06) | 4.86 (0.07)

19. Primary Outcome: Personal Motivation to Reduce Drug-related HIV-Risk Behavior (1-5)
Description: as for outcome 16
Time Frame: 6-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 95 | 90
units on a scale | 4.87 (0.06) | 4.78 (0.06)

20. Primary Outcome: Personal Motivation to Reduce Drug-related HIV-Risk Behavior (1-5)
Description: as for outcome 16
Time Frame: 12-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 95 | 90
units on a scale | 4.88 (0.04) | 4.92 (0.04)

21. Primary Outcome: Social Motivation to Reduce Drug-related HIV-Risk Behavior (1-5)
Description: Participants completed a questionnaire assessing their social motivation to reduce HIV risk behavior (e.g., "Most people who are important to me think I should always clean my needles before I share them with someone else during the next three months") and rated on a scale of 1 to 5, with higher scores indicating stronger social motivation to reduce HIV-risk behavior.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.65 (0.08) | 4.72 (0.09)

22. Primary Outcome: Social Motivation to Reduce Drug-related HIV-Risk Behavior (1-5)
Description: as for outcome 21
Time Frame: Immediately Post-Intervention, at 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.77 (0.08) | 4.69 (0.08)

23. Primary Outcome: Social Motivation to Reduce Drug-related HIV-Risk Behavior (1-5)
Description: as for outcome 21
Time Frame: 3-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.90 (0.04) | 4.85 (0.05)

24. Primary Outcome: Social Motivation to Reduce Drug-related HIV-Risk Behavior (1-5)
Description: as for outcome 21
Time Frame: 6-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.73 (0.07) | 4.91 (0.07)

25. Primary Outcome: Social Motivation to Reduce Drug-related HIV-Risk Behavior (1-5)
Description: as for outcome 21
Time Frame: 12-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.63 (0.09) | 4.75 (0.09)

26. Primary Outcome: Self-efficacy to Reduce Drug-related HIV-Risk Behavior (1-5)
Description: Participants completed a questionnaire assessing their self-efficacy about reducing HIV risk behavior (e.g., "How hard would it be for you to always use condoms") and rated on a scale of 1 to 5, with higher scores indicating greater self-efficacy to reduce HIV-risk behavior.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.01 (0.10) | 4.00 (0.11)

27. Primary Outcome: Self-efficacy to Reduce Drug-related HIV-Risk Behavior (1-5)
Description: as for outcome 26
Time Frame: Immediately Post-Intervention, at 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.41 (0.05) | 4.38 (0.09)

28. Primary Outcome: Self-efficacy to Reduce Drug-related HIV-Risk Behavior (1-5)
Description: as for outcome 26
Time Frame: 3-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.42 (0.08) | 4.36 (0.09)

29. Primary Outcome: Self-efficacy to Reduce Drug-related HIV-Risk Behavior (1-5)
Description: as for outcome 26
Time Frame: 6-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.22 (0.09) | 4.45 (0.10)

30. Primary Outcome: Self-efficacy to Reduce Drug-related HIV-Risk Behavior (1-5)
Description: as for outcome 26
Time Frame: 12-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.38 (0.08) | 4.52 (0.08)

31. Primary Outcome: Female Condom Skills (0-100%)
Description: Participants' HIV risk reduction behavioral skills were assessed based on the percentage of correct necessary steps demonstrated to properly select and apply a female condom using a replica.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: percentage of correct steps
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
percentage of correct steps | 57.60 (1.69) | 59.38 (1.78)

32. Primary Outcome: Female Condom Skills (0-100%)
Description: as for outcome 31
Time Frame: Immediately Post-Intervention, at 4 weeks
Measure: Mean (Standard Error); unit: percentage of correct steps
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
percentage of correct steps | 82.54 (1.25) | 74.32 (1.31)

33. Primary Outcome: Female Condom Skills (0-100%)
Description: as for outcome 31
Time Frame: 3-month follow up
Measure: Mean (Standard Error); unit: percentage of correct steps
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
percentage of correct steps | 79.29 (1.38) | 79.07 (1.45)

34. Primary Outcome: Female Condom Skills (0-100%)
Description: as for outcome 31
Time Frame: 6-month follow up
Measure: Mean (Standard Error); unit: percentage of correct steps
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
percentage of correct steps | 83.03 (1.19) | 80.86 (1.26)

35. Primary Outcome: Female Condom Skills (0-100%)
Description: as for outcome 31
Time Frame: 12-month follow up
Measure: Mean (Standard Error); unit: percentage of correct steps
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
percentage of correct steps | 83.37 (1.19) | 82.19 (1.25)

36. Primary Outcome: Male Condom Skills (0-100%)
Description: Participants' HIV risk reduction behavioral skills were assessed based on the percentage of correct necessary steps demonstrated to properly select and apply a male condom using a replica.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: percentage of correct steps
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
percentage of correct steps | 71.63 (1.35) | 73.97 (1.42)

37. Primary Outcome: Male Condom Skills (0-100%)
Description: as for outcome 36
Time Frame: Immediately Post-Intervention, at 4 weeks
Measure: Mean (Standard Error); unit: percentage of correct steps
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
percentage of correct steps | 87.23 (1.40) | 82.71 (1.47)

38. Primary Outcome: Male Condom Skills (0-100%)
Description: as for outcome 36
Time Frame: 3-month follow up
Measure: Mean (Standard Error); unit: percentage of correct steps
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
percentage of correct steps | 85.01 (1.22) | 84.64 (1.28)

39. Primary Outcome: Male Condom Skills (0-100%)
Description: as for outcome 36
Time Frame: 6-month follow up
Measure: Mean (Standard Error); unit: percentage of correct steps
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
percentage of correct steps | 87.51 (1.04) | 87.64 (1.09)

40. Primary Outcome: Male Condom Skills (0-100%)
Description: as for outcome 36
Time Frame: 12-month follow up
Measure: Mean (Standard Error); unit: percentage of correct steps
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
percentage of correct steps | 86.70 (1.17) | 85.95 (1.24)

41. Primary Outcome: Condom Use (0-4)
Description: Participants were asked: "In the past week, how much of the time did you use a condom or other latex protection when you had oral, anal, or vaginal sex?" and rated on scale of 0 to 4, with indicating greater condom use.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 3.80 (0.24) | 3.56 (0.26)

42. Primary Outcome: Condom Use (0-4)
Description: as for outcome 41
Time Frame: Immediately Post-Intervention, at 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 3.61 (0.24) | 3.56 (0.26)

43. Primary Outcome: Condom Use (0-4)
Description: as for outcome 41
Time Frame: 3-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 3.95 (0.24) | 3.75 (0.25)

44. Primary Outcome: Condom Use (0-4)
Description: as for outcome 41
Time Frame: 6-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 3.65 (0.24) | 3.79 (0.25)

45. Primary Outcome: Condom Use (0-4)
Description: as for outcome 41
Time Frame: 12-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 3.73 (0.24) | 3.83 (0.25)

46. Primary Outcome: Sex-related HIV-risk Reduction Knowledge (0-1)
Description: Participants' knowledge of sex-related HIV-risk reduction was assessed by being asked: "If an HIV positive person only has sex with another HIV positive person, they don't need to use condoms" and rated on a scale of 0 to 1, with a higher score indicating greater HIV-risk reduction knowledge.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 0.87 (0.03) | 0.91 (0.03)

47. Primary Outcome: Sex-related HIV-risk Reduction Knowledge (0-1)
Description: as for outcome 46
Time Frame: Immediately Post-Intervention, at 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 1.00 (0.02) | 0.95 (0.02)

48. Primary Outcome: Sex-related HIV-risk Reduction Knowledge (0-1)
Description: as for outcome 46
Time Frame: 3-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 0.97 (0.02) | 0.93 (0.02)

49. Primary Outcome: Sex-related HIV-risk Reduction Knowledge (0-1)
Description: as for outcome 46
Time Frame: 6-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 0.97 (0.02) | 0.95 (0.02)

50. Primary Outcome: Sex-related HIV-risk Reduction Knowledge (0-1)
Description: as for outcome 46
Time Frame: 12-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 0.98 (0.01) | 0.99 (0.01)

51. Primary Outcome: Personal Motivation to Reduce Sex-related HIV- Risk Behavior (1-5)
Description: Participants completed a questionnaire assessing their personal motivation to reduce sex-related HIV-risk behavior (e.g., "Always using condoms during sexual intercourse during the next three months would be good") and were rated on a scale of 1 to 5, with a higher score indicating greater personal motivation to reduce HIV-risk behavior.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.20 (0.09) | 4.26 (0.09)

52. Primary Outcome: Personal Motivation to Reduce Sex-related HIV- Risk Behavior (1-5)
Description: as for outcome 51
Time Frame: Immediately Post-Intervention, at 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.41 (0.08) | 4.24 (0.08)

53. Primary Outcome: Personal Motivation to Reduce Sex-related HIV- Risk Behavior (1-5)
Description: as for outcome 51
Time Frame: 3-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.39 (0.08) | 4.24 (0.09)

54. Primary Outcome: Personal Motivation to Reduce Sex-related HIV- Risk Behavior (1-5)
Description: as for outcome 51
Time Frame: 6-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.40 (0.08) | 4.29 (0.08)

55. Primary Outcome: Personal Motivation to Reduce Sex-related HIV- Risk Behavior (1-5)
Description: as for outcome 51
Time Frame: 12-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.21 (0.09) | 4.22 (0.09)

56. Primary Outcome: Social Motivation to Reduce Sex-related HIV- Risk Behavior (1-5)
Description: Participants completed a questionnaire assessing their social motivation to reduce sex-related HIV-risk behavior (e.g., "Most people who are important to me think I should always use condoms during sexual intercourse in the next three months") and were rated on a scale of 1 to 5, with a higher score indicating stronger social motivation to reduce HIV-risk behavior.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.67 (0.07) | 4.81 (0.08)

57. Primary Outcome: Social Motivation to Reduce Sex-related HIV- Risk Behavior (1-5)
Description: as for outcome 56
Time Frame: Immediately Post-Intervention, at 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.73 (0.07) | 4.75 (0.07)

58. Primary Outcome: Social Motivation to Reduce Sex-related HIV- Risk Behavior (1-5)
Description: as for outcome 56
Time Frame: 3-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.73 (0.07) | 4.71 (0.07)

59. Primary Outcome: Social Motivation to Reduce Sex-related HIV- Risk Behavior (1-5)
Description: as for outcome 56
Time Frame: 6-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.75 (0.07) | 4.77 (0.07)

60. Primary Outcome: Social Motivation to Reduce Sex-related HIV- Risk Behavior (1-5)
Description: as for outcome 56
Time Frame: 12-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.57 (0.08) | 4.70 (0.08)

61. Primary Outcome: Self-efficacy to Reduce Sex-related HIV- Risk Behavior (1-5)
Description: Participants completed a questionnaire assessing their self-efficacy about reducing sex-related HIV-risk behavior (e.g., "If asked, I am confident I could demonstrate how to use male condom and female condoms correctly") and were rated on a scale of 1 to 5, with a higher score indicating greater self-efficacy to reduce sex-related HIV-risk behavior.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 3.00 (0.12) | 3.09 (0.13)

62. Primary Outcome: Self-efficacy to Reduce Sex-related HIV- Risk Behavior (1-5)
Description: as for outcome 61
Time Frame: Immediately Post-Intervention, at 4 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 2.99 (0.12) | 3.06 (0.13)

63. Primary Outcome: Self-efficacy to Reduce Sex-related HIV- Risk Behavior (1-5)
Description: as for outcome 61
Time Frame: 3-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 3.02 (0.12) | 3.14 (0.12)

64. Primary Outcome: Self-efficacy to Reduce Sex-related HIV- Risk Behavior (1-5)
Description: as for outcome 61
Time Frame: 6-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.75 (0.07) | 4.77 (0.07)

65. Primary Outcome: Self-efficacy to Reduce Sex-related HIV- Risk Behavior (1-5)
Description: as for outcome 61
Time Frame: 12-month follow up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | CHRP Group | Control Condition
Number analyzed (Participants) | 97 | 92
units on a scale | 4.57 (0.08) | 4.70 (0.08)

ADVERSE EVENTS:
Time Frame: March 2007 through August 2011.
Arm/Group | CHRP Group | Control Condition
Serious Adverse Events (participants affected / at risk) | 0/149 | 0/155
Other Adverse Events (participants affected / at risk) | 0/149 | 0/155

LIMITATIONS AND CAVEATS:
The drug-risk reducing effects of methadone may have restricted our ability to detect intervention effects on drug-related outcomes. Participants may have also been reluctant to report HIV risk related behaviors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes